CLINICAL TRIAL: NCT07248397
Title: Development and Validation of a Screening Tool for Preschool Children Aged 1-6 Years
Status: Active, not recruiting | Type: Observational
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 202401410B0
Record Dates: First submitted 2025-11-18; First posted 2025-11-25 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-09

CONDITIONS: Early Childhood Development (ECD)
Keywords: Chatbot-Assisted Developmental Assessment Scale for Preschool Children (CADAS); preschool children; motor development; cognitive development; language development; social-emotional development

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Preschool Children: Children aged 1-6 years enrolled in preschools and nurseries in Taoyuan City.
  Interventions: Other: No Intervention: Observational Cohort

INTERVENTIONS:
Other: No Intervention: Observational Cohort — This is an observational study. No intervention or treatment is administered. Participants complete developmental assessments for research purposes only.

SUMMARY:
This study develops and validates the Chatbot-Assisted Developmental Assessment Scale for Preschool Children (CADAS), a screening tool for 1-6-year-olds. Using AI and the Kebbi Air S robot, CADAS assesses motor, cognitive, language, and social-emotional development through interactive games. A total of 180 children will participate, comparing AI-robot and human assessments for reliability and validity. The project aims to create a localized, efficient, and accurate developmental screening tool to support early detection and improve child development services in Taiwan.

DETAILED DESCRIPTION:
Current developmental assessments in Taiwan rely mainly on foreign tools, which limit cultural suitability. This study addresses that gap by creating a local, AI-based screening system using Kebbi Air S, a social robot capable of voice prompts, facial recognition, and data recording. Five game-like scenarios will assess different developmental domains; one will be robot-assisted and four human-administered for comparison. 180 children (1-6 years) will be recruited from a nonprofit preschool in Taoyuan, with 60 also taking the Comprehensive Developmental Inventory for Infants and Toddlers (CDIIT) for validation. Analyses using SPSS 21.0 and ConQuest 4.5 will test reliability, validity, and item quality. The study aims to build a reliable local tool and confirm the feasibility of chatbot-assisted evaluation, contributing to a national preschool development database and improving early intervention accuracy.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 1-6 years enrolled in preschools or nurseries in Taoyuan City.
* Parent or guardian consent obtained.
* Able to follow basic instructions and complete play-based tasks

Exclusion Criteria:

* Diagnosed developmental, neurological, or genetic disorders.
* Severe visual, hearing, or motor impairments affecting task performance.
* No parental consent or early withdrawal during assessment.

Ages: 1 Year to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Preschool children from Taoyuan City, Taiwan.
Sampling Method: Non-Probability Sample
Enrollment: 180 (Estimated)
Dates: Start 2024-09-23 (Actual); Primary Completion 2027-09-22 (Estimated); Study Completion 2027-09-22 (Estimated)

PRIMARY OUTCOMES:
Motor Development Score | Baseline
  Motor score from CADAS, manually administered by trained research assistants to assess gross and fine motor skills through play-based tasks.
Cognitive Development Score | Baseline
  Cognitive score from CADAS, assessed manually through structured play evaluating reasoning, attention, and memory.
Language Development Score | Baseline
  Language score from CADAS, obtained from human-administered tasks testing receptive and expressive language.
Social-Emotional Development Score | Baseline
  Social-emotional score from Scenario 3 using the Kebbi Air S robot. Robot-guided prompts and facial recognition are used to assess emotion and interaction, compared with manual ratings.

CONTACTS AND LOCATIONS:
Overall Officials: Chia-Ling Chen, Study Director — Chang Gung Memorial Hospital
Locations (1):
- Chang Gung Memorial Hospital, Taoyuan District, Taiwan